CLINICAL TRIAL: NCT05963711
Title: The Penile Microbiome in Partners of Women with Recurrent BV and Its Response to Decolonization Protocol
Brief Title: The Genital Microbiome of Male Partners of Women with Recurrent BV Undergoing Vaginal Microbiome Transplantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Ahinoam Lev-Sagie, Professor, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0463-22-HMO
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Bacterial Vaginosis; Microbial Colonization
Keywords: Penile microbiome; Vaginal microbiome transplant; Male partners; Bacterial vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: In those with BV-associated penile microbiome, a decolonization attempt will be conducted, (daily wash for 5 days with chlorhexidine gluconate 4%). if decolonization fails, an antibiotic cream will be used to eradicate BV associated bacteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: chlorhexidine gluconate 4% — In case BV associated bacteria will be identified (using molecular sequencing) in male samples, decolonization attempt will be conducted, using a daily wash for 5 days with chlorhexidine gluconate 4%. Following decolonization attempt, male participants will undergo re- sampling, to assess for microbiome changes.
  In case there is no change in microbial composition, partners will be instructed to repeat decolonization protocol, and apply a 2 cm diameter volume of 2% clindamycin cream topically to the head of the penis and upper shaft (under the foreskin if uncircumcised) twice daily for seven days following repeated decolonization. Re-sampling will follow.
  Other Names: 2% clindamycin cream

SUMMARY:
There is strong observational evidence that sexual activity plays a key role in Bacterial Vaginosis (BV) acquisition and recurrence. Microbiological data support the contribution of sexual transmission to the pathogenesis of BV through the exchange of BV-associated bacteria (BVAB) between sexual partners.

Although BV epidemiology strongly suggests sexual transmission, treatment of sexual partners is not recommended, based on prior treatment studies of male partners of women with recurrent BV, which showed no benefit with male treatment. Nevertheless, male condom use is highly protective against recurrent BV.

This study aims to evaluate the male-partner's genital microbiome as a potential source of BV-recurrence in women undergoing vaginal microbiota transplantation (NCT04517487), and whether disinfection can eliminate BV-associated penile microbiome.

ELIGIBILITY:
Inclusion Criteria:

* The subject has s female partner who participates in VMT study ( NCT04517487).
* The subject is defined by the woman as her male regular partner.
* Willing to use a condom as instructed by the protocol.
* Willing to comply with decolonization protocol.

Exclusion Criteria:

* A known skin disease involving the penile skin.
* A known sensitivity to chlorhexidine gluconate
* Any of the partners (female/male) has more than one sexual partner.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Penile microbiome composition | 1 year
  Characterization of the penile microbial communities using shotgun analysis, and their similarity to the vaginal microbiota composition of their sexual partner.
Penile microbiome composition after disinfection | 1 year
  Characterization of the penile microbiome composition using shotgun analysis, after disinfection protocol or antibiotic use.

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No